CLINICAL TRIAL: NCT05549661
Title: Phase 1 Study to Determine the Safety and Efficacy of Onvansertib, A Novel, Oral, PLK1 Inhibitor in Patients With Proliferative Chronic Myelomonocytic Leukemia (CMML) and Myelodysplastic Syndrome/MPN Overlap Neoplasms Relapsed/Refractory or Intolerant to Available Therapies
Brief Title: Onvansertib for the Treatment of Recurrent or Refractory Chronic Myelomonocytic Leukemia and Myelodysplastic Syndrome/MPN Overlap Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210807; NCI-2022-07695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA272496 (NIH); 22-005600 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Chronic Myelomonocytic Leukemia; Refractory Chronic Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Not Otherwise Specified; Recurrent Atypical Chronic Myeloid Leukemia; Recurrent Myelodysplastic/Myeloproliferative Neoplasm; Refractory Myelodysplastic/Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myelodysplastic-Myeloproliferative Diseases | interventions — Specimen Handling; Biopsy; onvansertib; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (onvansertib) (Experimental): Patients receive onvansertib PO QD on study. Patients also undergo bone marrow aspiration and biopsy, collection of blood samples, and ultrasound imaging during screening and throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Onvansertib; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Onvansertib — Given PO
  Other Names: 'PLK1 Inhibitor PCM-075; NMS-1286937; PCM 075; PCM-075; PLK-1 Inhibitor PCM-075; Polo-like Kinase 1 Inhibitor NMS-1286937; Polo-like Kinase 1 Inhibitor PCM-075
Procedure: Ultrasound Imaging — Undergo ultrasound imaging
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase I trial evaluates the safety, effectiveness, and best dose of onvansertib for the treatment of patients with chronic myelomonocytic leukemia and Myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) overlap neoplasms that has come back (recurrent) or that does not respond to treatment (refractory). Onvansertib is a drug that binds to and inhibits an enzyme called PLK1, preventing cancer cell proliferation and causing cell death.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterization of adverse events (AEs) by type, incidence, severity [graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0], seriousness, and relationship to treatment; effects on vital signs and laboratory parameters; changes from baseline in electrocardiograms (ECGs), physical examinations, weight, and Eastern Cooperative Oncology Group (ECOG) performance status.

SECONDARY OBJECTIVES:

I. Efficacy: complete response (CR) rate, according to the 2015 myelodysplastic syndrome (MDS)/myeloproliferative neoplasm (MPN) International Working Group (IWG) criteria.

II. Overall remission rate (ORR), defined as CR + complete cytogenetic remission + partial remission (CR+ complete cytogenetic remission [CCR] + partial remission [PR]).

III. Volumetric spleen response rate, as determined by ultrasound scan (US). IV. Constitutional symptoms, as assessed by the MPN-Symptom Assessment Form (SAF) total symptom score (TSS).

EXPLORATORY OBJECTIVES:

I. Onvansertib activity in RAS mutant subtypes of proliferative chronic myelomonocytic leukemia (CMML).

II. Monocyte subset analysis by flow cytometry (CD14/CD16). III. Relation of genomic backgrounds and changes, as assessed by next generation sequencing (NGS), to response.

IV. Relation between changes in mutant circulating-tumor deoxyribonucleic acid (ctDNA) and response.

V. CR rate, ORR and spleen response rate as per the 2015 MDS/MPN IWG response criteria.

VI. Assessment of target engagement. VII. Expression levels of PLK1 and KMT2A.

OUTLINE: This is a dose-escalation study of onvansertib followed by a dose-expansion study.

Patients receive onvansertib orally (PO) once daily (QD) on study. Patients also undergo bone marrow aspiration and biopsy, collection of blood samples, and ultrasound imaging during screening and throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION - INCLUSION CRITERIA:

* Age >= 18 years
* History of World Health Organization (WHO)-defined diagnosis of proliferative CMML (WBC count >= 13,000/mm^3 at time of diagnosis), or MDS/MPN overlap neoplasm with WBC count >= 13,000/mm3 at time of diagnosis (atypical CML and MDS/MPN-NOS).

  * NOTE: Hydroxyurea or hypomethylating induced leukopenia does not preclude inclusion. Discussion of WBC < 13,000/mm^3 due to treatment at the time of preregistration must be discussed with the Sponsor/Principal Investigator
* Relapsed/refractory following treatment with hydroxyurea; or at least 4 cycles of treatment with hypomethylating agents; or who are intolerant of treatment with either therapy. Note: Prior exposure to erythropoiesis stimulating agents is allowed. Hydroxyurea may continue for the first 28 days on study. Continuation of hydroxyurea beyond the first cycle must be discussed with the Sponsor/Principal Investigator
* Willing and able to review, understand, and provide written consent before starting any study-specific procedures or therapy
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory bone marrow specimens for correlative research
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Recovered to grade 1 or baseline or established as sequelae from all toxic effects of previous therapy except alopecia
* Platelet count >= 20,000/mm^3 (obtained =< 14 days prior to pre-registration)

  * NOTE: For platelet count < 20,000/mm3 and in situations where the primary investigator deems the thrombocytopenia to be attributable to the underlying CMML, patients can be enrolled as long as they are able to achieve a platelet count of 20,000/mm3 with transfusional support
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (=< 3 x ULN for patients with Gilbert's syndrome) (obtained =< 14 days prior to pre-registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (obtained =< 14 days prior to pre-registration)
* Estimated glomerular filtration rate (eGFR) >= 50 mL/min/m^2 using one of the following methods (obtained =< 14 days prior to pre-registration):

  * Chronic Kidney Disease-Epidemiology Collaboration (CKDEPI) 2021 formula
  * Corrected creatinine clearance via serum and 24-hour urine creatinine assessment
  * Iothalamate/Iohexol glomerular filtrate rate via plasma/urine assessment
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research

REGISTRATION - INCLUSION CRITERIA:

* Histological confirmation of WHO-defined diagnosis of a myelodysplastic/myeloproliferative neoplasm (MDS/MPN) including one of the following (NOTE: to confirm patient is still eligible and has not progressed to

AML):

* Proliferative CMML
* Atypical chronic myeoloid leukemia (aCML)
* MDS/MPN not otherwise specified (MDS/MPN, NOS)
* NOTE: Hydroxyurea or hypomethylating agent induced leukopenia does not preclude inclusion. Discussion of WBC < 13,000/mm^3 due to treatment at the time of registration must be discussed with the Sponsor/Principal Investigator.

  * For a man or a woman of child-bearing potential (WOCBP): Must agree to use contraception or take measures to avoid pregnancy during the study and for 180 days after the final dose of any study drug. Adequate contraception is defined as follows:
* Complete true abstinence
* Consistent and correct use of one of the following methods of birth control:

  * Male partner who is sterile prior to the female patient's entry into the study and is the sole sexual partner for that female patient
  * Implants of levonorgestrel
  * Injectable progestogen
  * Intrauterine device (IUD) with a documented failure rate of less than 1% per year
  * Oral contraceptive pill (either combined or progesterone only)
  * Barrier method, for example: diaphragm with spermicide or condom with spermicide in combination with either implants of levonorgestrel or injectable progestogen

    * WOCBP must have a negative serum or urine pregnancy test =< 7 days prior to registration
* NOTE: WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months); or women on hormone replacement therapy with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an IUD or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (eg, vasectomy), must be considered to be of child-bearing potential
* NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria:

PRE-REGISTRATION - EXCLUSION CRITERIA:

* Previous exposure to an alternative (investigational) PLK1 inhibitor
* Demonstration of transformation to acute leukemia on any prior bone marrow biopsy
* Prior allogeneic hematopoietic stem cell transplantation with active grade 2-4 graft-versus-host disease (GVHD) or with moderate to severe chronic GVHD

  * NOTE: The patient should not have received calcineurin inhibitors ≤28 days prior to pre-registration and should not be actively receiving immunosuppressive therapy for acute or chronic GVHD.
  * NOTE: CMML or MDS/MPN overlap neoplasms relapse after allogeneic stem cell transplant is allowed as long as they are >100 days after transplant and do not have the aforementioned GVHD criteria.
* Active central nervous system disease
* Concurrent active malignancy, except adequately treated nonmelanoma skin cancer. History of curatively treated in situ cancer of the cervix, curatively treated in situ cancer of the breast, or other solid tumors curatively treated is allowed as long as there is no evidence of disease for > 2 years

  * NOTE: Precursor states such as monoclonal gammopathy of undetermined significance (MGUS), monoclonal B-cell lymphocytosis (MBL), and indolent lymphoproliferative disorders must be discussed with the Sponsor/Principal Investigator.
* New York Heart Association (NYHA) class III/IV heart failure or active angina/angina equivalents
* Anticancer chemotherapy (exception: hydroxyurea) or biologic therapy administered within 2 weeks (and at least 4 elimination half-lives for clinical trial agents) prior to pre-registration. NOTE: Hydroxyurea is allowed for the first 28 days on study. Continuation of hydroxyurea beyond the first cycle must be discussed with the Sponsor/Principal Investigator
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Major surgery =< 6 weeks prior to pre-registration
* Gastrointestinal (GI) disorder(s) that, in the opinion of the Investigator, would significantly impede the absorption of an oral agent (eg, intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection)
* Unable or unwilling to swallow study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant nonhealing or healing wounds, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Known active infection with human immunodeficiency virus (HIV) with measurable viral titer, hepatitis B surface antigen positivity, or hepatitis C with measurable viral titer. NOTE: Patients with antibody to hepatitis B core antibody are eligible if they have no measurable viral titer. Patients who have had a hepatitis B virus (HBV) immunization are eligible
* Patient is receiving any live vaccine (eg, varicella, pneumococcus) =< 28 days prior to pre-registration. NOTE: messenger ribonucleic acid (mRNA)-based (eg, Pfizer or Moderna) or replication-deficient virus (eg, Oxford/AstraZeneca) COVID19 vaccines are permitted
* Disease requiring systemic treatment with systemic immunosuppression with steroid steroids at a dose of >= 20 mg/day prednisone (or equivalent). Exceptions: Intermittent use of bronchodilators or inhaled steroids, local steroid injections, topical steroids
* Any active disease condition that would render the protocol treatment dangerous or impair the ability of the patient to receive study drug
* Strong CYP3A4 inhibitors/inducers as identified per institutional guidelines
* QT interval with Fridericia's correction (QTcF) > 470 milliseconds. In the case of potentially correctible causes of QT prolongation, (eg, medications, hypokalemia), the electrocardiogram (ECG) may be repeated once during screening and that result may be used to determine eligibility

REGISTRATION - EXCLUSION CRITERIA:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Increased risk of Torsade des Pointes (TdP) defined as follows:

  * A marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval > 480 msec [CTCAE Grade >= 2] using Fredericia's QT correction formula)
  * A history of additional risk factors for TdP (eg. heart failure, family history of long QT syndrome)
* Transformation to acute leukemia on registration bone marrow biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 4 years
  Safety will be assessed primarily based on reported adverse events (AEs). The severity of AEs will be graded as mild, moderate, severe, or life-threatening according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All reported toxicities, regardless of attribution, will be summarized by toxicity type and maximum grade, and sorted by number of patients experiencing the toxicity. The maximum grade consolidates the reports of a given toxicity for a patient over time by taking the maximum across time.

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 4 years
  CR will be determined by the International Working Group (IWG) response criteria. CR rate will be presented descriptively for each cohort, with 95% confidence intervals (CIs).
Overall remission rate (ORR) | Up to 4 years
  ORR is defined as CR + complete cytogenetic remission + partial response and will be determined by the IWG response criteria. ORR will be presented descriptively for each cohort, with 95% CIs.
Volumetric spleen response | Up to 4 years
  Spleen volumes, as determined by ultrasound, will be summarized descriptively for each cohort.
Constitutional symptoms | Up to 4 years
  The Myeloproliferative Neoplasm-Symptom Assessment Form total symptom score will be summarized descriptively for each cohort. Symptom scores will also be summarized individually.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal S. Patnaik, MBBS, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials